CLINICAL TRIAL: NCT01604408
Title: A Phase 2 Randomized Study to Investigate the Efficacy and Safety of LY2495655 Versus Placebo in Older Patients Who Have Fallen Recently and Have Muscle Weakness
Brief Title: A Study in Older Participants Who Have Fallen and Have Muscle Weakness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14499; I1Q-MC-JDDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — landogrozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2495655 (Experimental): Participants received a 315-milligram (mg) dose of LY2495655, administered subcutaneously (SC), every 4 weeks (Q4W) for 20 weeks.
  Interventions: Biological: LY2495655
- Placebo (Placebo Comparator): Participants received a LY2495655-matching dose of placebo, administered SC, Q4W for 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: LY2495655 — Administered SC
  Arms: LY2495655
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
LY2495655 is an investigational drug being tested for muscle wasting.

ELIGIBILITY:
Inclusion Criteria:

* Sustained at least 1 fall within 1 calendar year before study screening.
* Requires ≥12 seconds to perform a repeated chair stands test or is unable to complete this test at screening.
* Hand grip strength is ≤37 kilograms (kg) for men (81.4 pounds) or ≤21 kg for women (46.2 pounds) at screening.
* Can stand up from a chair and walk ≥10 meters without human assistance (gait aids such as cane[s], crutches, or walkers are acceptable) at screening.
* Able to climb at least 1 step on a staircase without human assistance according to the participant at screening (using handrails is allowed).
* Have screening clinical laboratory test results within normal reference range for the population, or have results with acceptable deviations that are judged to be not clinically significant by the investigator.

Exclusion Criteria:

* Major lower limb pain or neurologic impairment or vestibular vertigo or visual impairment that could severely confound measures of physical performance.
* Recent lower limb fracture and/or major lower limb surgery.
* Planned major surgical procedure within 6 months following study drug dosing.
* Have had a lower extremity amputation of the foot, leg, and/or thigh.
* Have a body mass index (BMI) ≥35 kilogram per meter squared (kg/m2).
* Severe vitamin D deficiency.
* Underlying muscle disease other than age-associated muscle waste or disuse atrophy.
* Current use or previous use of any drugs known to influence muscle mass or performance.
* Have had a recent neurologic injury (<6 months before study drug dosing), such as stroke or spinal cord injury.
* History of a malignant neoplasm in the 18 months before first study drug dosing.
* Have a history or presence of unstable cardiovascular or pulmonary comorbidities.
* Have a positive fecal occult blood (FOB) test at screening, or the participant cannot provide a stool sample for FOB testing before first study drug dosing.
* Have either severe ongoing liver disease or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 times upper limit of normal (ULN), alkaline phosphatase (ALP) >1.5 times ULN, or total bilirubin >1.5 times ULN at screening.
* Have an estimated creatinine clearance <20 milliliters per minute (mL/minute).
* Have a history of severe allergic reaction to a monoclonal antibody.
* Are males with a female partner of childbearing potential who do not agree to use contraception during the treatment period of the study and up to 15 weeks after the last dose of investigational product (study drug).
* Have known allergies to LY2495655, its constituents, or related compounds.
* Have severe active psychiatric disease or cognitive impairment as assessed by the Mini-Mental State Examination (MMSE) score <22 (for a participant who went to school up to age 15 years or less) or <24 (for a participant who went to school up to at least age 16), making the participant unlikely to understand the informed consent form or comply with protocol procedures.
* Exhibit excessive consumption of alcohol or abuse of drugs.
* Have uncontrolled diabetes mellitus.
* Have had ocular trauma, ophthalmologic surgery, or eye laser treatment within 6 months before study drug dosing.
* Have hyponatremia (serum sodium levels <135 millimoles/liter ([mmol/L]) at screening unless a retest shows normonatremia before study drug dosing.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galveston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hornsby, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingswood, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daw Park, South Australia
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pierre-Bénite
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuttgart
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huddinge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mölndal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala

REFERENCES:
- [Derived] Becker C, Lord SR, Studenski SA, Warden SJ, Fielding RA, Recknor CP, Hochberg MC, Ferrari SL, Blain H, Binder EF, Rolland Y, Poiraudeau S, Benson CT, Myers SL, Hu L, Ahmad QI, Pacuch KR, Gomez EV, Benichou O; STEADY Group. Myostatin antibody (LY2495655) in older weak fallers: a proof-of-concept, randomised, phase 2 trial. Lancet Diabetes Endocrinol. 2015 Dec;3(12):948-57. doi: 10.1016/S2213-8587(15)00298-3. Epub 2015 Oct 27. PMID 26516121

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | LY2495655 | Placebo
Started | 102 | 99
Received at Least 1 Dose of Study Drug | 102 | 99
Completed | 102 | 98
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Treatment Period 2
Arm/Group | LY2495655 | Placebo
Started | 102 | 98
Completed | 100 | 96
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 3
Arm/Group | LY2495655 | Placebo
Started | 100 | 96
Completed | 95 | 91
Not Completed | 5 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Sponsor Decision | 1 | 0
Period: Treatment Period 4
Arm/Group | LY2495655 | Placebo
Started | 95 | 91
Completed | 92 | 89
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 5
Arm/Group | LY2495655 | Placebo
Started | 92 | 89
Completed | 88 | 89
Not Completed | 4 | 0
Not completed — Adverse Event | 4 | 0
Period: Treatment Period 6
Arm/Group | LY2495655 | Placebo
Started | 88 | 89
Completed | 86 | 87
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Sponsor decision | 0 | 1
Period: Observation Period
Arm/Group | LY2495655 | Placebo
Started | 86 | 87
Completed | 85 | 84
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study.
Groups:
- LY2495655: Participants received a 315-mg dose of LY2495655, administered SC, Q4W for 20 weeks.
- Total: Total of all reporting groups
Arm/Group | LY2495655 | Placebo | Total
Number analyzed (Participants) | 102 | 99 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.84 (4.73) | 82.57 (5.20) | 82.20 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 65 | 140
  Male | 27 | 34 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 19 | 36
  Not Hispanic or Latino | 48 | 45 | 93
  Unknown or Not Reported | 37 | 35 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 101 | 98 | 199
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  France | 13 | 12 | 25
  United States | 37 | 36 | 73
  Argentina | 17 | 19 | 36
  Australia | 19 | 17 | 36
  Germany | 6 | 7 | 13
  Sweden | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Week Endpoint in Appendicular Lean Body Mass (aLBM)
Description: Change from baseline to 24-week endpoint in aLBM, as measured by dual energy x-ray absorptiometry (DEXA), is presented. Least squares (LS) means were calculated using a mixed model repeated measures (MMRM) with treatment, visit, and treatment-by-visit interaction as fixed effects and baseline aLBM as covariate.
Time Frame: Baseline to 24 weeks
Population: All participants who received at least 1 dose of LY2495655 or placebo with evaluable aLBM data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2495655 | Placebo
Number analyzed (Participants) | 77 | 82
kilograms (kg) | 0.303 (0.085) | -0.123 (0.083)
Statistical Analysis 1: Comparison: LY2495655 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean Difference = 0.426, 95% CI 2-sided [0.192 to 0.660]

2. Secondary Outcome: Change From Baseline in Stair Climbing (StC) Time
Description: Change from baseline to the 24-week endpoint in StC time is presented. StC time was assessed by measuring the fastest time achieved to climb 4 steps on a 4-step staircase (the test was performed 2 times). LS means were calculated using a MMRM with treatment, visit, and treatment-by-visit interaction as fixed effects and baseline StC score as covariate.
Time Frame: Baseline to 24 weeks
Population: All participants who received at least 1 dose of LY2495655 or placebo with evaluable StC time data.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | LY2495655 | Placebo
Number analyzed (Participants) | 80 | 84
seconds | -0.276 (0.182) | 0.184 (0.178)
Statistical Analysis 1: Comparison: LY2495655 vs Placebo; Test type: Superiority or Other; p = 0.073, Mixed Model Repeated Measures; LS Mean Difference = -0.461, 90% CI 2-sided [-0.883 to -0.039]

3. Secondary Outcome: Change From Baseline in Repeated Chair Stands (RCS) Time
Description: Change from baseline to 24-week endpoint in RCS time is presented. In the RCS test, participants were asked to rise from a chair 5 times as fast as possible with their arms folded on their chest. Performance was measured in seconds, as the time from the initial seated position to the final standing position. LS means were calculated using an MMRM with treatment, visit, and treatment-by-visit interaction as fixed effects and baseline RCS time as covariate.
Time Frame: Baseline to 24 weeks
Population: All participants who received at least 1 dose of LY2495655 or placebo with evaluable RCS time data.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | LY2495655 | Placebo
Number analyzed (Participants) | 53 | 64
seconds | -1.888 (0.588) | 0.826 (0.551)
Statistical Analysis 1: Comparison: LY2495655 vs Placebo; Test type: Superiority or Other; p = 0.191, Mixed Model Repeated Measures; LS Mean Difference = -1.062, 90% CI 2-sided [-2.400 to 0.276]

4. Secondary Outcome: Change From Baseline in Usual Gait Speed (uGS) at 4 Meters
Description: Change from baseline to the 24-week endpoint in uGS is presented. Two attempts to walk a 4-meter distance were made. LS means were calculated using a MMRM with treatment, visit, and treatment-by-visit interaction as fixed effects and baseline uGS as covariate.
Time Frame: Baseline to 24 weeks
Population: All participants who received at least 1 dose of LY2495655 or placebo with evaluable uGS data.
Measure: Least Squares Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | LY2495655 | Placebo
Number analyzed (Participants) | 80 | 85
meters per second (m/s) | 0.030 (0.017) | 0.013 (0.017)
Statistical Analysis 1: Comparison: LY2495655 vs Placebo; Test type: Superiority or Other; p = 0.478, Mixed Model Repeated Measures; LS Mean Difference = 0.017, 90% CI 2-sided [-0.023 to 0.057]

ADVERSE EVENTS:
Arm/Group | LY2495655 | Placebo
Serious Adverse Events (participants affected / at risk) | 27/102 | 18/99
Other Adverse Events (participants affected / at risk) | 90/102 | 77/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2495655 (N=102) | Placebo (N=99)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth socket haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2495655 (N=102) | Placebo (N=99)
Constipation (Gastrointestinal disorders) | 7 (8) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 7 (8)
Asthenia (General disorders) | 4 (4) | 5 (5)
Fatigue (General disorders) | 12 (14) | 3 (3)
Injection site bruising (General disorders) | 6 (8) | 0 (0)
Injection site pain (General disorders) | 20 (69) | 5 (7)
Pain (General disorders) | 5 (5) | 6 (8)
Nasopharyngitis (Infections and infestations) | 7 (10) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 7 (9) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (9) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9) | 10 (10)
Headache (Nervous system disorders) | 7 (8) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days